CLINICAL TRIAL: NCT02468791
Title: A Randomized, Double-blind, Parallel-group Comparative Bioequivalence Trial of MabionCD20® (Mabion SA) Compared to MabThera® (Rituximab, Roche) in Patients With Rheumatoid Arthritis
Brief Title: MabionCD20® Compared to MabThera® in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mabion SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MabionCD20-001RA
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Autoimmune Diseases; Rituximab; Immune System Diseases; Joint Diseases; Rheumatic Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases; Immune System Diseases; Joint Diseases; Rheumatic Diseases | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MabionCD20® (Experimental): A course of MabionCD20® in rheumatoid arthritis patients consists of two 1000 mg intravenous infusions with two weeks interval.
  Interventions: Drug: Rituximab
- MabThera® (Active Comparator): A course of MabThera® (Rituximab, Roche) in rheumatoid arthritis patients consists of two 1000 mg intravenous infusions with two weeks interval.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
The purpose of this study is to evaluate biosimilarity between test product MabionCD20® and the reference product - MabThera® (rituximab) and to demonstrate comparative safety and tolerability of a single course of treatment of MabionCD20® and MabThera® in patients with moderate to severe active rheumatoid arthritis.

DETAILED DESCRIPTION:
Subjects who meet the criteria for participation in this study receive 2 intravenous infusions of MabionCD20® or MabThera® with two weeks interval in combination with methotrexate and folic acid. After the treatment period, patients are followed for 24 weeks, in order to continue checking safety. Therefore, the total study lasts 48 weeks. There is a possibility to repeat treatment after 6 months of the first infusions if subject meets the retreatment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis with disease duration minimum 6 months prior to screening visit
* Patients who are naive to tumor necrosis factor (TNF) antagonists or any other monoclonal antibody therapies
* Patients who have had an inadequate response to an adequate regimen of methotrexate

Exclusion Criteria:

* History of current rheumatic autoimmune disease other than RA and current inflammatory joint disease other than RA
* Contraindications according to the MabThera SmPC and every serious coexisting diseases which, in the Investigator's opinion, would preclude subject participation
* Positive tests for HIV, hepatitis B surface antigen (HBsAg) Anti-HBc antibody, hepatitis C antibody
* Prior treatment with rituximab, other anti-CD20 mAb, anti-TNF-alpha drug or any other monoclonal antibodies
* Pregnancy or lactation or women planning to get pregnant during the course of the study and/or within 12 months post last study drug infusion
* Allergic reaction or intolerance to rituximab, MabionCD20 or any of their components
* Severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or previous treatment of any lymphocyte-depleting therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in each treatment group achieving the primary efficacy endpoint of a ≥ 20% improvement on the American College of Rheumatology score (ACR20) at Week 24. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (51):
- Bosnia and Herzegovina (5):
  - Clinical Centre Banja Luka Location Paprikovac, Banja Luka
  - University Clinical Hospital Mostar, Mostar
  - Clinical Centre University of Sarajevo, Sarajevo
  - General Hospital "Dr. Abdulah Nakas", Sarajevo
  - University Clinical Centre Tuzla, Tuzla
- Georgia (7):
  - Carabs Medline Ltd, Tbilisi
  - Cardio-Reanimation Center Ltd, Tbilisi
  - Diagnostic Service ltd, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - MediClub Georgia, Tbilisi
  - Medicore Ltd, Tbilisi
  - Medulla-Chemotherapy and Immunotherapy Clinic, Tbilisi
- Poland (23):
  - Centrum Miriada, Bialystok
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Położnicze św Łukasza Sp.z.o.o, Częstochowa
  - NSZOZ Unica CR, Dopiewo
  - Wojewódzki Szpital Zespolony, Elblag
  - Małopolskie Centrum Medyczne S.C., Krakow
  - Szpital Uniwersytecki, Oddział Kliniczny Kliniki Chorób Wewnętrznych, Krakow
  - Szpital Specjalistyczny im. J. Dietla, Krakow
  - Ośrodek Badań Klinicznych, Lublin
  - REUMED, Lublin
  - NZOZ Lecznica MAK-MED. S.C., Nadarzyn
  - Centrum Medyczne Nowa Sól, Nowa Sól
  - SOLUMED, Poznan
  - AL Klinika, Poznan
  - NZOZ Poradnia Leczenia Osteoporozy i Chorób Narządu Ruchu, Stalowa Wola
  - Zespół Opieki Zdrowotnej w Suchej Beskidzkiej, Sucha Beskidzka
  - Śląski Szpital Reumatologiczo-Rehabilitacyjny im. Generała Jerzego Ziętka, Ustroń
  - Linea Corporis Spółka z Ograniczoną Odpowiedzialnością, Warsaw
  - IRMED, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - Medica Pro Familia Sp. z o.o. S.K.A, Warsaw
  - Instytut Reumatologii, Warsaw
  - KO-MED Centra Kliniczne, Zamość
- Serbia (4):
  - Institute for Rheumatology - Belgrade, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Institute for treatment and rehabilitation "Niska Banja", Niška Banja
  - Clinical center of Vojvodina, Clinic for medical rehabilitation, Novi Sad
- Ukraine (12):
  - Communal Medical Institution "City Clinical Hospital no 3", Chernivtsi
  - National Medical University, Chair of Internal Medicine based on Ivano-Frankivsk Central Clinical City Hospital, Ivano-Frankivsk
  - Department of Cardiology and Functional Diagnostics, Kharkiv Medical Academy of Postgraduated Education, Kharkiv
  - Kharkiv City Clinical Hospital no 27, Kharkiv
  - Regional Hospital Veterans of War, Kharkiv
  - State Institute "L T Malaya Institute of Therapy of NAMS of Ukraine", Kharkiv
  - Administration of Medical Service and Rehabilitation of "ARTEM" State Holding Company, Kyiv
  - National Scientific Center "M.D. STRAZHESKO INSTITUTE OF CARDIOLOGY, MAS OF UKRAINE", Kyiv
  - Chair of Internal Medicine no 2 of Ternopil State Medical University, Ternopil
  - Uzhgorod Clinical Hospital of the Lviv Railways, Department of Therapy, Uzhhorod
  - Clinical City Hospital no 7, Zaporizhzhia
  - Zaporizhzhia Medical Academy of Postgraduate Education of Ministry of Health of Ukraine, Zaporizhzhia